CLINICAL TRIAL: NCT06828185
Title: Patient Reported Experiences With Sparing ExteRnal Oblique Fascia Vs Standard Inguinal OrchiEctomy
Acronym: PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5250002
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Testicular Cancer
Keywords: orchiectomy; postoperative pain; testis cancer; germ cell tumors
MeSH Terms: conditions — Testicular Neoplasms; Pain, Postoperative; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical inguinal orchiectomy (Active Comparator)
  Interventions: Procedure: Radical inguinal orchiectomy
- Radical external oblique fascia sparing orchiectomy (Active Comparator)
  Interventions: Procedure: Radical external oblique fascia sparing orchiectomy

INTERVENTIONS:
Procedure: Radical inguinal orchiectomy — External oblique fascia will be incised during orchiectomy
  Arms: Radical inguinal orchiectomy
Procedure: Radical external oblique fascia sparing orchiectomy — External oblique fascia will be spared during orchiectomy
  Arms: Radical external oblique fascia sparing orchiectomy

SUMMARY:
The purpose of this study is to evaluate the difference in patient-reported postoperative outcomes between two standard-of-care surgical techniques for radical orchiectomy (inguinal orchiectomy versus external oblique fascia sparing orchiectomy) for treatment of patients with suspected testicular malignancy. The main questions it aims to answer are:

1. Does sparing the external oblique fascia during orchiectomy reduce pain after surgery?
2. Is there a difference in narcotic consumption after surgery?
3. Is there a difference in neuropathic pain after surgery?
4. Is there a difference in complications after surgery?

DETAILED DESCRIPTION:
Radical inguinal orchiectomy is the standard of care surgical approach for removing a testicle when clinically there is concern for testicular cancer. The procedure is generally minor and performed in the outpatient setting. Recent data demonstrates a trend towards high opioid prescription following this procedure in an attempt to minimize postoperative pain, which is associated with persistent new opioid use in the future. Numerous efforts have been put in place to minimize postoperative pain following scrotal procedures, with success noted when opioid sparing pathways have been adopted. However, there has been sparse data on modifications within surgical technique that could improve patient pain following this procedure.

There have been various descriptions of technique to performing a radical orchiectomy which involves removal of the diseased testicle and spermatic cord. Classically, performing a radical inguinal orchiectomy involves incision of the external oblique fascia to expose and ligate the spermatic cord. During this step, the ilioinguinal nerve is exposed and can be injured by either traction injury or inadvertent transection. Modifications to this technique have been described which involve sparing of the external oblique fascia. Both approaches are performed via a similar incision and both the testicle and spermatic cord are removed. In fascia sparing modification, the spermatic cord is controlled, dissected, and subsequently ligated at the level of the superficial inguinal ring without incising the external oblique fascia. Proponents of this approach suggest the potential for less convalescence and faster recovery due to less tissue manipulation and avoidance of disturbances to the ilioinguinal nerve. Despite this potential benefit, there is no evidence to demonstrate superiority of either approach as it relates to patient recovery.

Therefore, we propose a randomized single-blinded clinical trial investigating postoperative pain outcomes of inguinal radical orchiectomy compared to external oblique fascia sparing radical orchiectomy.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing radical orchiectomy for suspected testicular malignancy
* Testicular malignancy can be germ cell tumor or non germ cell tumors, including paratesticular tumors as long as a radical orchiectomy is planned
* Participants over 18 years of age who can provide informed consent
* Participants not currently using opiates for another reason
* Regional and metastatic patients are allowed, as long as participant does not require opiates for pain related to metastatic disease
* No contraindication for participant to receive standardized medication pathway in the peri-operative period.

Exclusion Criteria:

* Clinical T4 disease
* History of illicit substance abuse (including prior opioid abuse) except for marijuana
* Participants who underwent chemotherapy or radiotherapy prior to orchiectomy
* Opioid use within 1 month of study enrollment
* Participants with large testis masses requiring skin incision larger than 8 cm in size.
* Participants with large testis masses requiring orchiectomy through an incision other than the standard transverse inguinal incision (i.e. hockey stick incision, vertical incision)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Level | Change between Postoperative day 0 [the day surgery was completed] through postoperative day 7
  Post-operative pain levels will be measured by the Short Form Inguinal Pain Score (sf-IPQ) The score range is between 0 and 12, with zero points indicating no pain and 12 points indicating the most intense pain. Scores for subjects undergoing inguinal orchiectomy will be compared to subjects undergoing external oblique fascia sparing radical orchiectomy.

SECONDARY OUTCOMES:
Opioid consumption | Change between Postoperative day 0 [the day surgery was completed] through postoperative day 7
  Subjects will self-report the total number of Oxycodone 5 mg tablets consumed for breakthrough pain during the first post-op week. There is no pre-defined range for this self-report but the higher the number of tablets consumed may be an indication of great pain intensity.
Neuropathic Pain Level | Change between Postoperative day 0 [the day surgery was completed] through postoperative day 7)
  Post-Operative Neuropathic pain levels will be measured by the modified Barrow Neurological Institute hypesthesia scale. A total score ranging between 1 and 4, with 1 representing minimal neuropathic pain and 4 representing intense neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shei A, Rice JB, Kirson NY, Bodnar K, Birnbaum HG, Holly P, Ben-Joseph R. Sources of prescription opioids among diagnosed opioid abusers. Curr Med Res Opin. 2015 Apr;31(4):779-84. doi: 10.1185/03007995.2015.1016607. Epub 2015 Feb 24. PMID 25661018